CLINICAL TRIAL: NCT00140205
Title: Pharmacokinetics of Leptin Administration During Fasting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Christos Mantzoros, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2001P000260
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2017-05

CONDITIONS: Energy Deficiency Due to Short-term Fasting
Keywords: leptin; fasting; pharmacokinetics
MeSH Terms: conditions — Fasting | interventions — recombinant methionyl human leptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fed state or fasting state (Experimental): 1-day fed studies with administration of r-metHuLeptin at three different doses (0.01 mg/kg, 0.1 mg/kg, 0.3 mg/kg). All subjects participated in 3 studies in the fed condition (Part A) and 3 separate 72-hour fasting studies.
  Intervention administered was-r-metreleptin in 3 different doses
  Interventions: Drug: r-metHuLeptin

INTERVENTIONS:
Drug: r-metHuLeptin — r-metreleptin was given in 3 different dose in fed and fasting states
  Other Names: Recombinant leptin

SUMMARY:
The purpose of this study will be to determine the correct dose of leptin, a natural hormone secreted by the fat cells, to give to people when they are fasting and also to determine whether giving leptin to a person when he or she is fasting will reverse the changes in hormone levels that occur with fasting.

DETAILED DESCRIPTION:
Leptin is a newly-identified hormone secreted by fat cells under normal conditions that acts in the brain to decrease appetite and increase long term energy usage. Leptin levels usually go down when people are not eating for extended periods of time. Changes in metabolism and certain hormone levels also occur with fasting. By studying the pharmacokinetics of leptin administration, we can evaluate the changes of leptin levels in response to giving different doses of leptin as well as acute changes of other hormones in response to leptin levels. Investigations such as this one have important implications for the future therapeutic use of leptin, including determining the appropriate dose of leptin to use in future studies involving leptin administration.

Comparison: subjects receiving leptin at 3 different doses in the fed state compared to the fasting state

ELIGIBILITY:
Inclusion Criteria:

* healthy men with body mass indices (BMI) <25 kg/m2)
* overweight otherwise healthy men with BMI > 27 kg/m2
* healthy lean women with BMI<25 kg/m2
* overweight otherwise healthy women with BMI > 27 kg/m2

Exclusion Criteria:

* history of any illness that may affect the concentrations of the hormones that will be studied (such as anemia, infectious diseases, renal or hepatic failure, diabetes mellitus, cancer, lymphoma, hypogonadism, malabsorption or malnourishment, hypo or hyperthyroidism, hypercortisolism, alcoholism or drug abuse, eating disorders)
* on medications known to affect the hormones to be measured in this study (such as glucocorticoids, anti-seizure medications or thyroid hormones)
* known history of anaphylaxis or anaphylactoid-like reactions or who have a known hypersensitivity to E. Coli derived proteins
* women who are breast feeding, pregnant, or wanting to become pregnant during the next 6 months

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2001-02; Primary Completion 2004-06 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos S Mantzoros, MD DSc FACP FACE, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Bouzoni E, Perakakis N, Connelly MA, Angelidi AM, Pilitsi E, Farr O, Stefanakis K, Mantzoros CS. PCSK9 and ANGPTL3 levels correlate with hyperlipidemia in HIV-lipoatrophy, are regulated by fasting and are not affected by leptin administered in physiologic or pharmacologic doses. Metabolism. 2022 Sep;134:155265. doi: 10.1016/j.metabol.2022.155265. Epub 2022 Jul 9. PMID 35820631
- [Derived] Chrysafi P, Perakakis N, Farr OM, Stefanakis K, Peradze N, Sala-Vila A, Mantzoros CS. Leptin alters energy intake and fat mass but not energy expenditure in lean subjects. Nat Commun. 2020 Oct 13;11(1):5145. doi: 10.1038/s41467-020-18885-9. PMID 33051459
- [Derived] Moragianni VA, Aronis KN, Chamberland JP, Mantzoros CS. Short-term energy deprivation alters activin a and follistatin but not inhibin B levels of lean healthy women in a leptin-independent manner. J Clin Endocrinol Metab. 2011 Dec;96(12):3750-8. doi: 10.1210/jc.2011-1453. Epub 2011 Sep 14. PMID 21917874
- [Derived] Aronis KN, Diakopoulos KN, Fiorenza CG, Chamberland JP, Mantzoros CS. Leptin administered in physiological or pharmacological doses does not regulate circulating angiogenesis factors in humans. Diabetologia. 2011 Sep;54(9):2358-67. doi: 10.1007/s00125-011-2201-x. Epub 2011 Jun 10. PMID 21660636
- [Derived] Scheer FA, Chan JL, Fargnoli J, Chamberland J, Arampatzi K, Shea SA, Blackburn GL, Mantzoros CS. Day/night variations of high-molecular-weight adiponectin and lipocalin-2 in healthy men studied under fed and fasted conditions. Diabetologia. 2010 Nov;53(11):2401-5. doi: 10.1007/s00125-010-1869-7. Epub 2010 Aug 12. PMID 20703446
- See also: Click here for more information about the Mantzoros Research Group. — http://www.bidmc.org/Research/Departments/Medicine/Divisions/Endocrinology/Laboratories/MantzorosLab.aspx
- See also: Click here for more information about Beth Israel Deaconess Medical Center. — http://www.bidmc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- 5 LEAN MEN Fasting State (72 Hrs) on 0.3mg/kg Leptin: 5 lean men were fasted for 72 hrs and during that period recieved 0.3mg/kg leptin
- 5 OBESE MEN 72 HR FASTING on 0.3mg/kg Leptin: 5 obese men were fasted for 72 hrs and during that period received 0.3mg/kg leptin
- 5 LEAN WOMEN 72 HR FATSING on 0.3mg/kg Leptin: 5 lean women were fasted for 72 hrs and during that period received 0.3mg/kg leptin
Period: Overall Study
Arm/Group | 5 LEAN MEN Fasting State (72 Hrs) on 0.3mg/kg Leptin | 5 OBESE MEN 72 HR FASTING on 0.3mg/kg Leptin | 5 LEAN WOMEN 72 HR FATSING on 0.3mg/kg Leptin
Started | 5 | 5 | 5
Completed | 5 | 5 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- LEAN MEN 24h Fed or 72h Fasting in Different Leptin Doses: 5 lean men were fasted for 72 hrs and during that period received 0.01 mg/kg leptin (First visit), 0,1 mg/kg (Second visit), 0.3 mg/kg (Third visit)
- OBESE MEN 24h Fed or 72h Fasting in Different Leptin Doses: 5 obese men were fasted for 72 hrs and during that period recieved 0.01 mg/kg leptin (First visit), 0,1 mg/kg (Second visit), 0.3 mg/kg (Third visit)
- OBESE WOMEN 24h Fed or 72h Fasting in Different Leptin Doses: 5 lean women were fasted for 72 hrs and during that period received 0.01 mg/kg leptin (First visit), 0,1 mg/kg (Second visit), 0.3 mg/kg (Third visit)
- Total: Total of all reporting groups
Arm/Group | LEAN MEN 24h Fed or 72h Fasting in Different Leptin Doses | OBESE MEN 24h Fed or 72h Fasting in Different Leptin Doses | OBESE WOMEN 24h Fed or 72h Fasting in Different Leptin Doses | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 5 | 15
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 22 (.09) | 23 (.08) | 22 (.05) | 23 (.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 5 | 5
  Male | 5 | 5 | 0 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 5 | 15
BMI [Number; unit: participants]
  BMI>30kg/m2 | 0 | 5 | 0 | 5
  BMI<25kg/m2 | 5 | 0 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Leptin Pharmacokinetic Parameters - TIME(T1/2) DAY 3 / TMAX DAY 3 72-hour Fasting Day 3 Leptin Dose 0.01 mg/kg
Description: 72-hour fasting Day 3 Leptin dose 0.01 mg/kg
Time Frame: 3 DAY
Measure: Mean (Standard Deviation); unit: HR
Arm/Group | 5 LEAN MEN Fasting (72 Hrs) - Leptin 0.01 mg/kg | 5 OBESE MEN Fasting (72 Hrs) - Leptin 0.01 mg/kg | 5 LEAN WOMEN Fasting (72 Hrs) - Leptin 0.01 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
HR
  TIME(T1/2) DAY 3 | 1.93 (0.28) | 2.75 (1.49) | 2.99 (1.01)
  TMAX DAY 3 | 2.00 (0.71) | 3.00 (0.71) | 2.80 (1.30)

2. Primary Outcome: Leptin Pharmacokinetics Parameters - c(MAX) / L0 (ENDOGENOUS LEPTIN LEVEL) 72-hour Fasting Day 3 Leptin Dose 0.01 mg/kg
Description: 72-hour fasting Day 3 Leptin dose 0.01 mg/kg
Time Frame: 3 DAY
Measure: Mean (Standard Deviation); unit: NG/ML
Arm/Group | 5 LEAN MEN Fasting State (72 Hrs) | 5 OBESE MEN 72 HR FASTING | 5 LEAN WOMEN 72 HR FATSING
Number analyzed (Participants) | 5 | 5 | 5
NG/ML
  c(MAX) | 2.60 (0.59) | 4.21 (1.17) | 4.62 (1.60)
  L0 (ENDOGENOUS LEPTIN LEVEL) | 1.42 (0.72) | 3.32 (1.21) | 3.53 (1.26)

3. Primary Outcome: Leptin Pharmacokinetics Parameters - AUC 72-hour Fasting Day 3 Leptin Dose 0.01 mg/kg
Description: 72-hour fasting Day 3 Leptin dose 0.01 mg/kg
Time Frame: 3 DAY
Measure: Mean (Standard Deviation); unit: NG*H/ML
Arm/Group | 5 LEAN MEN Fasting State (72 Hrs) | 5 OBESE MEN 72 HR FASTING | 5 LEAN WOMEN 72 HR FATSING
Number analyzed (Participants) | 5 | 5 | 5
NG*H/ML | 12.27 (2.95) | 35.43 (13.81) | 47.81 (23.90)

4. Primary Outcome: Leptin Pharmacokinetic Parameters TIME(T1/2) DAY 3 / TMAX DAY 3 72-hour Fasting Day 3 Leptin Dose 0.1 mg/kg
Description: 72-hour fasting Day 3 Leptin dose 0.1 mg/kg
Time Frame: 3 DAY
Measure: Mean (Standard Deviation); unit: HR
Arm/Group | 5 LEAN MEN Fasting (72 Hrs) - Leptin 0.1 mg/kg | 5 OBESE MEN Fasting (72 Hrs) - Leptin 0.1 mg/kg | 5 LEAN WOMEN (72 Hrs) Fasting - Leptin 0.1 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
HR
  TIME(T1/2) DAY 3 | 1.82 (0.58) | 3.10 (1.20) | 1.73 (0.57)
  TMAX DAY 3 | 3.20 (1.10) | 4.00 (1.58) | 3.00 (1.00)

5. Primary Outcome: Leptin Pharmacokinetics Parameters - c(MAX) / L0 (ENDOGENOUS LEPTIN LEVEL) 72-hour Fasting Day 3 Leptin Dose 0.1 mg/kg
Description: 72-hour fasting Day 3 Leptin dose 0.1 mg/kg
Time Frame: 3 DAY
Measure: Mean (Standard Deviation); unit: NG/ML
Arm/Group | 5 LEAN MEN Fasting State (72 Hrs) - Leptin 0.1 mg/kg | 5 OBESE MEN Fasting (72 Hrs) - Leptin 0.1 mg/kg | 5 LEAN WOMEN Fasting (72 Hrs)- Leptin 0.1 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
NG/ML
  c(MAX) | 33.88 (9.38) | 78.43 (14.71) | 106.4 (36.7)
  L0 (ENDOGENOUS LEPTIN LEVEL) | 1.69 (0.89) | 5.92 (1.33) | 5.36 (1.89)

6. Primary Outcome: Leptin Pharmacokinetics Parameters - AUC 72-hour Fasting Day 3 Leptin Dose 0.1 mg/kg
Description: 72-hour fasting Day 3 Leptin dose 0.1 mg/kg
Time Frame: 3 DAY
Measure: Mean (Standard Deviation); unit: NG*H/ML
Arm/Group | 5 LEAN MEN Fasting State (72 Hrs) - Leptin 0.1 mg/kg | 5 OBESE MEN Fasting (72 Hrs) - Leptin 0.1 mg/kg | 5 LEAN WOMEN Fasting (72 Hrs)- Leptin 0.1 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
NG*H/ML | 206.9 (56.9) | 778.2 (121.5) | 676.5 (267.4)

7. Primary Outcome: Leptin Pharmacokinetic Parameters - TIME(T1/2) DAY 3 / TMAX DAY 3 72-hour Fasting Day 3 Leptin Dose 0.3 mg/kg
Description: 72-hour fasting Day 3 Leptin dose 0.3 mg/kg
Time Frame: 3 DAY
Measure: Mean (Standard Deviation); unit: HR
Arm/Group | 5 LEAN MEN Fasting (72 Hrs) - Leptin 0.3 mg/kg | 5 OBESE MEN Fasting (72 Hrs) - Leptin 0.3 mg/kg | 5 LEAN WOMEN Fasting (72 Hrs)- Leptin 0.3 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
HR
  TIME(T1/2) DAY 3 | 1.98 (0.28) | 2.40 (0.54) | 1.92 (0.45)
  TMAX DAY 3 | 3.80 (1.30) | 3.40 (1.67) | 3.80 (1.48)

8. Primary Outcome: Leptin Pharmacokinetics Parameters - c(MAX) / L0 (ENDOGENOUS LEPTIN LEVEL) 72-hour Fasting Day 3 Leptin Dose 0.3 mg/kg
Description: 72-hour fasting Day 3 Leptin dose 0.3 mg/kg
Time Frame: 3 DAY
Measure: Mean (Standard Deviation); unit: NG/ML
Arm/Group | 5 LEAN MEN Fasting (72 Hrs) - Leptin 0.3 mg/kg | 5 OBESE MEN Fasting (72 Hrs) - Leptin 0.3 mg/kg | 5 LEAN WOMEN Fasting (72 Hrs)- Leptin 0.3 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
NG/ML
  c(MAX) | 88.39 (32.13) | 301.6 (86.8) | 399.6 (76.8)
  L0 (ENDOGENOUS LEPTIN LEVEL) | 1.62 (0.64) | 13.72 (2.97) | 6.95 (1.05)

9. Primary Outcome: Leptin Pharmacokinetics Parameters - AUC 72-hour Fasting Day 3 Leptin Dose 0.3 mg/kg
Description: 72-hour fasting Day 3 Leptin dose 0.3 mg/kg
Time Frame: 3 DAY
Measure: Mean (Standard Deviation); unit: NG*H/ML
Arm/Group | 5 LEAN MEN Fasting (72 Hrs) - Leptin 0.3 mg/kg | 5 OBESE MEN Fasting (72 Hrs) - Leptin 0.3 mg/kg | 5 LEAN WOMEN Fasting (72 Hrs)- Leptin 0.3 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
NG*H/ML | 747.3 (300.8) | 2717 (647.1) | 2738 (624)

10. Primary Outcome: Leptin Pharmacokinetic Parameters - TIME(T1/2) / TMAX 24-hour Fed Leptin Dose 0.3 mg/kg
Description: 24-hour fed Leptin dose 0.3 mg/kg
Time Frame: 1 DAY
Measure: Mean (Standard Deviation); unit: HR
Arm/Group | 5 LEAN MEN Fed (24 Hrs) - Leptin 0.3 mg/kg | 5 OBESE MEN Fed (24 Hrs) - Leptin 0.3 mg/kg | 5 LEAN WOMEN Fed (24 Hrs) - Leptin 0.3 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
HR
  TIME(T1/2) | 2.94 (0.95) | 3.69 (1.13) | 2.91 (0.90)
  TMAX | 3.60 (0.89) | 3.40 (1.67) | 2.80 (0.84)

11. Primary Outcome: Leptin Pharmacokinetics Parameters - c(MAX) / L0 (ENDOGENOUS LEPTIN LEVEL) 24-hour Fed Leptin Dose 0.3 mg/kg
Description: 24-hour fed Leptin dose 0.3 mg/kg
Time Frame: 1 DAY
Measure: Mean (Standard Deviation); unit: NG/ML
Arm/Group | 5 LEAN MEN Fed (24 Hrs) - Leptin 0.3 mg/kg | 5 OBESE MEN Fed (24 Hrs) - Leptin 0.3 mg/kg | 5 LEAN WOMEN Fed (24 Hrs) - Leptin 0.3 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
NG/ML
  c(MAX) | 168.7 (61.7) | 254.3 (36.7) | 440.7 (85.2)
  L0 (ENDOGENOUS LEPTIN LEVEL) | 2.97 (0.68) | 16.24 (5.00) | 12.60 (7.78)

12. Primary Outcome: Leptin Pharmacokinetics Parameters - AUC 24-hour Fed Leptin Dose 0.3 mg/kg
Description: 24-hour fed Leptin dose 0.3 mg/kg
Time Frame: 1 DAY
Measure: Mean (Standard Deviation); unit: NG*H/ML
Arm/Group | 5 LEAN MEN Fed (24 Hrs) - Leptin 0.3 mg/kg | 5 OBESE MEN Fed (24 Hrs) - Leptin 0.3 mg/kg | 5 LEAN WOMEN Fed (24 Hrs) - Leptin 0.3 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
NG*H/ML | 1243 (304.2) | 2948 (521.9) | 3300 (871)

13. Primary Outcome: Leptin Pharmacokinetic Parameters - TIME(T1/2) / TMAX 24-hour Fed Leptin Dose 0.01 mg/kg
Description: 24-hour fed Leptin dose 0.01 mg/kg
Time Frame: 1 DAY
Measure: Mean (Standard Deviation); unit: HR
Arm/Group | 5 LEAN MEN Fed (24 Hrs) - Leptin 0.01 mg/kg | 5 OBESE MEN Fed (24 Hrs) - Leptin 0.01 mg/kg | 5 LEAN WOMEN Fed (24 Hrs) - Leptin 0.01 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
HR
  TIME(T1/2) | 2.84 (0.98) | 4.71 (2.16) | 3.08 (1.24)
  TMAX | 3.00 (1.00) | 6.20 (3.35) | 2.80 (0.84)

14. Primary Outcome: Leptin Pharmacokinetics Parameters - c(MAX) / L0 (ENDOGENOUS LEPTIN LEVEL) 24-hour Fed Leptin Dose 0.01 mg/kg
Description: 24-hour fed Leptin dose 0.01 mg/kg
Time Frame: 1 DAY
Measure: Mean (Standard Deviation); unit: NG/ML
Arm/Group | 5 LEAN MEN Fed (24 Hrs) - Leptin 0.01 mg/kg | 5 OBESE MEN Fed (24 Hrs) - Leptin 0.01 mg/kg | 5 LEAN WOMEN Fed (24 Hrs) - Leptin 0.01 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
NG/ML
  c(MAX) | 5.97 (1.65) | 7.91 (2.37) | 14.51 (2.96)
  L0 (ENDOGENOUS LEPTIN LEVEL) | 2.32 (0.48) | 12.67 (6.15) | 15.54 (8.90)

15. Primary Outcome: Leptin Pharmacokinetics Parameters - AUC 24-hour Fed Leptin Dose 0.01 mg/kg
Description: 24-hour fed Leptin dose 0.01 mg/kg
Time Frame: 1 DAY
Measure: Mean (Standard Deviation); unit: NG*H/ML
Arm/Group | 5 LEAN MEN Fed (24 Hrs) - Leptin 0.01 mg/kg | 5 OBESE MEN Fed (24 Hrs) - Leptin 0.01 mg/kg | 5 LEAN WOMEN Fed (24 Hrs) - Leptin 0.01 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
NG*H/ML | 33.18 (8.68) | 113.9 (56.6) | 110.5 (45.0)

16. Primary Outcome: Leptin Pharmacokinetic Parameters - TIME(T1/2) / TMAX 24-hour Fed Leptin Dose 0.1 mg/kg
Description: 24-hour fed Leptin dose 0.1 mg/kg
Time Frame: 1 DAY
Measure: Mean (Standard Deviation); unit: HR
Arm/Group | 5 LEAN MEN Fed (24 Hrs) - Leptin 0.1 mg/kg | 5 OBESE MEN Fed (24 Hrs) - Leptin 0.1 mg/kg | 5 LEAN WOMEN Fed (24 Hrs) - Leptin 0.1 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
HR
  TIME(T1/2) | 2.89 (0.24) | 4.72 (1.51) | 2.08 (1.01)
  TMAX | 3.00 (1.58) | 4.60 (0.89) | 3.20 (0.84)

17. Primary Outcome: Leptin Pharmacokinetics Parameters - c(MAX) / L0 (ENDOGENOUS LEPTIN LEVEL) 24-hour Fed Leptin Dose 0.1 mg/kg
Description: 24-hour fed Leptin dose 0.1 mg/kg
Time Frame: 1 DAY
Measure: Mean (Standard Deviation); unit: NG/ML
Arm/Group | 5 LEAN MEN Fed (24 Hrs) - Leptin 0.1 mg/kg | 5 OBESE MEN Fed (24 Hrs) - Leptin 0.1 mg/kg | 5 LEAN WOMEN Fed (24 Hrs) - Leptin 0.1 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
NG/ML
  c(MAX) | 72.56 (12.19) | 77.26 (10.10) | 107.4 (19.4)
  L0 (ENDOGENOUS LEPTIN LEVEL) | 2.11 (0.50) | 15.49 (8.64) | 14.36 (11.12)

18. Primary Outcome: Leptin Pharmacokinetics Parameters - AUC 24-hour Fed Leptin Dose 0.1 mg/kg
Description: 24-hour fed Leptin dose 0.1 mg/kg
Time Frame: 1 DAY
Measure: Mean (Standard Deviation); unit: NG*H/ML
Arm/Group | 5 LEAN MEN Fed (24 Hrs) - Leptin 0.1 mg/kg | 5 OBESE MEN Fed (24 Hrs) - Leptin 0.1 mg/kg | 5 LEAN WOMEN Fed (24 Hrs) - Leptin 0.1 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
NG*H/ML | 507.4 (44.1) | 1051 (202.9) | 620.2 (157.1)

19. Secondary Outcome: Cytokine Levels 24h Fed or 72h Fasting for All Different Leptin Doses (0,01-0,1-0,3 mg/kg)
Description: Data were collected neither in Fed nor in Fasting state for the different doses of leptin
Time Frame: 1 DAY or DAY 3
Arm/Group | 5 LEAN MEN Fed (24h) or Fasting (72 Hrs) | 5 OBESE MEN Fed (24h) or Fasting (72 Hrs) | 5 LEAN WOMEN Fed (24h) or Fasting (72 Hrs)
Number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: Neuroendocrine Hormone Levels 24h Fed or 72h Fasting for All Different Leptin Doses (0,01-0,1-0,3 mg/kg)
Description: Data were collected neither in Fed nor in Fasting state for the different doses of leptin
Time Frame: 1 DAY or DAY 3
Arm/Group | 5 LEAN MEN Fed (24h) or Fasting (72 Hrs) | 5 OBESE MEN Fed (24h) or Fasting (72 Hrs) | 5 LEAN WOMEN Fed (24h) or Fasting (72 Hrs)
Number analyzed (Participants) | 0 | 0 | 0

21. Secondary Outcome: Adipokine Hormone Levels 24h Fed or 72h Fasting for All Different Leptin Doses (0,01-0,1-0,3 mg/kg)
Description: Data were collected neither in Fed nor in Fasting state for the different doses of leptin
Time Frame: day 3 of fasting and day 1 of fed state
Arm/Group | 5 LEAN MEN Fed (24h) or Fasting (72 Hrs) | 5 OBESE MEN Fed (24h) or Fasting (72 Hrs) | 5 LEAN WOMEN Fed (24h) or Fasting (72 Hrs)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Fasting State (72 Hrs)
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
small size population, results cannot be generalized

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No